CLINICAL TRIAL: NCT03708705
Title: Liquid Biopsy-based Monitoring System for Relapse of Hepatocellular Carcinoma Associated With Hepatitis B After Liver Transplantation: A Multi-center and Prospective Study
Brief Title: Liquid Biopsy-based Monitoring System for Relapse of HCC After Liver Transplantation: A Multi-center and Prospective Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Xiao Xu, professor, Zhejiang University
Other Study IDs: ZJUXU1177
Record Dates: First submitted 2018-10-13; First posted 2018-10-17 (Actual); Last update posted 2018-10-19 (Actual); Status verified 2018-10

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood and tissue samples.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Relapse: Relapse of tumor within two years after liver transplantation
  Interventions: Other: Risk model of tumor relapse
- Non-relapse: Non-relapse of tumor within two years after liver transplantation
  Interventions: Other: Risk model of tumor relapse

INTERVENTIONS:
Other: Risk model of tumor relapse — High risk factor model of tumor relapse after liver transplantation
  Other Names: Risk model

SUMMARY:
This study aims to develop a novel, reliable, liquid biopsy-based biomarker system for relapse of HCC associated with hepatitis B after liver transplantation.

DETAILED DESCRIPTION:
Relapse of hepatocellular carcinoma (HCC) is one of the leading causes of death after liver transplantation (LT). Detection of cancer at an earlier stage of the disease can be critical to improve patient survival. Liquid biopsy is a revolutionary technique that is opening previously unexpected perspectives. It consists of circulating extracellular vesicles, nucleic acids (DNA and RNA) and circulating tumor cells. The detection and isolation of circulating tumor cells, circulating tumor DNA and exosomes, as a source of genomic and proteomic information in patients with cancer. Regarding these promising and potential transformative tools, as well as the issues still needed to be addressed for adopting various liquid biopsy approaches into clinical practice. This study aims to develop a novel, reliable, liquid biopsy-based biomarker system for relapse of HCC associated with hepatitis B after liver transplantation.

ELIGIBILITY:
Inclusion Criteria:

transplants for HCC

Exclusion Criteria:

Liver transplantation due to other disease

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: hospitalization patients
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2018-11-20 (Estimated); Primary Completion 2020-05-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
relapse rate of tumor | two years

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR, Analytic Code
Time Frame: Two years